CLINICAL TRIAL: NCT05756881
Title: A Randomised Double-blind Placebo-controlled Study on the Effects of Topical Palm Tocotrienols on Blemish-prone Skin
Brief Title: Topical Palm Tocotrienols on Blemish-prone Skin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrawal
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Malaysia Palm Oil Board (Other Government); Avantsar Sdn. Bhd. (Unknown)
Responsible Party: Principal Investigator, Goh Choon Fu, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MA-T3-T3
Record Dates: First submitted 2023-02-10; First posted 2023-03-06 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Acne
Keywords: tocotrienol; acne; topical; skin
MeSH Terms: conditions — Acne Vulgaris | interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum containing 1.5 % w/w of palm-oil derived vitamin E concentrate (Active Comparator): Serum containing 1.5 % w/w of palm-oil derived vitamin E concentrate
  Interventions: Other: Cosmetic product
- Serum (placebo) (Placebo Comparator): Serum (placebo)
  Interventions: Other: Cosmetic product

INTERVENTIONS:
Other: Cosmetic product — Apply on the face twice a day

SUMMARY:
A single-center, double-blind, randomised, placebo-controlled parallel-group study.

Selected subjects will be randomised into active and control groups in a ratio of 1:1. Investigational products assigned will be applied on the facial skin as part of daily skin care routine. The effects will be observed during the 12-weeks of use.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy individuals, aged 18 years and above
2. Fitzpatrick skin type II to IV
3. Blemish-prone skin with acne of severity grade 2 or 3 based on Comprehensive Acne Severity Scale (CASS)

Exclusion Criteria:

1. Has a history of chronic drug or alcohol abuse
2. Is a current smoker
3. History of severe allergic reactions to topical products or vitamin E
4. Participant with severe and uncontrollable comorbidities (including but not limited to e.g. diabetes, hypertension, kidney failure)
5. Pregnant, breastfeeding, or planning pregnancy
6. Participant with known skin conditions (including but not limited to e.g. sensitive skin, eczema and diseased skin e.g. contact dermatitis), uncontrolled medical conditions, or any other condition that could interfere with the study evaluations or increase risk to the participant (such as polycystic ovary syndrome and contact dermatitis)
7. Participant with compromised/broken skin, tattoos, scarring, excessive hair growth, very uneven skin tone, or other conditions that would interfere with evaluations or increase risk
8. Participation in another study within 4 weeks of screening visit
9. Has severe acne or acne conglobata
10. Use of systemic treatment for acne such as isotretinoin, contraceptive pills, or spironolactone within 4 weeks of screening visit
11. Use of topical treatments like antibiotics, corticosteroids, benzoyl peroxide, azelaic acid, salicylic acid, alpha hydroxy acids (AHAs), vitamins A (retinol) or C (ascorbic acid) or their analogs or derivatives and other anti-inflammatory drugs within 2 weeks of screening visit
12. Use of scrub, alpha-hydroxy acid (AHA), skin irritant products in the 2 days before study treatment start
13. Participant with active bacterial/fungal/viral skin infections or susceptibility to such infections within 2 weeks of Screening visit
14. Use oral antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with at least 50% reduction in numbers of acne lesion or at least 2 grade improvement according to CASS from baseline | 18 Week
  Acne lesion count

SECONDARY OUTCOMES:
The percent change from baseline in global face total lesion count. | 18 Week
  Acne lesion count
Acne lesion counts for the total global face and total lesion counts | 18 Week
  Acne lesion count
CASS assessment | 18 Week
  Comprehensive Acne Severity Scale (CASS)
Survey (CADI) | 18 Week
  The Cardiff Acne Disability Index 2021
The percent change from baseline in sebum, skin pH, hydration and erythema index | 18 Week
  Skin probe

CONTACTS AND LOCATIONS:
Overall Officials: Choon Fu Goh, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- School of Pharmaceutical Sciences, Universiti Sains Malaysia, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sen CK, Khanna S, Roy S. Tocotrienols in health and disease: the other half of the natural vitamin E family. Mol Aspects Med. 2007 Oct-Dec;28(5-6):692-728. doi: 10.1016/j.mam.2007.03.001. Epub 2007 Mar 27. PMID 17507086
- [Background] Patel V, Rink C, Gordillo GM, Khanna S, Gnyawali U, Roy S, Shneker B, Ganesh K, Phillips G, More JL, Sarkar A, Kirkpatrick R, Elkhammas EA, Klatte E, Miller M, Firstenberg MS, Chiocca EA, Nesaretnam K, Sen CK. Oral tocotrienols are transported to human tissues and delay the progression of the model for end-stage liver disease score in patients. J Nutr. 2012 Mar;142(3):513-9. doi: 10.3945/jn.111.151902. Epub 2012 Feb 1. PMID 22298568
- [Background] Ikeda S, Niwa T, Yamashita K. Selective uptake of dietary tocotrienols into rat skin. J Nutr Sci Vitaminol (Tokyo). 2000 Jun;46(3):141-3. doi: 10.3177/jnsv.46.141. PMID 10955281
- [Background] Traber MG, Podda M, Weber C, Thiele J, Rallis M, Packer L. Diet-derived and topically applied tocotrienols accumulate in skin and protect the tissue against ultraviolet light-induced oxidative stress. Asia Pac J Clin Nutr. 1997 Mar;6(1):63-7. PMID 24394657
- [Background] Suzuki YJ, Tsuchiya M, Wassall SR, Choo YM, Govil G, Kagan VE, Packer L. Structural and dynamic membrane properties of alpha-tocopherol and alpha-tocotrienol: implication to the molecular mechanism of their antioxidant potency. Biochemistry. 1993 Oct 12;32(40):10692-9. doi: 10.1021/bi00091a020. PMID 8399214
- [Background] Thiele JJ, Traber MG, Podda M, Tsang K, Cross CE, Packer L. Ozone depletes tocopherols and tocotrienols topically applied to murine skin. FEBS Lett. 1997 Jan 20;401(2-3):167-70. doi: 10.1016/s0014-5793(96)01463-9. PMID 9013880
- [Background] Thiele JJ, Traber MG, Tsang K, Cross CE, Packer L. In vivo exposure to ozone depletes vitamins C and E and induces lipid peroxidation in epidermal layers of murine skin. Free Radic Biol Med. 1997;23(3):385-91. doi: 10.1016/s0891-5849(96)00617-x. PMID 9214574
- [Background] N.Z. Yusuf, Z.A. Azizul Hasan, R. Ismail, TOCOGELS As Anti-Inflammatory Agents, in: MPOB Information Series, Malaysian Palm Oil Board, Kuala Lumpur, Malaysia, 2011.
- [Background] Zouboulis CC. Acne and sebaceous gland function. Clin Dermatol. 2004 Sep-Oct;22(5):360-6. doi: 10.1016/j.clindermatol.2004.03.004. PMID 15556719
- [Background] Suppiah TSS, Sundram TKM, Tan ESS, Lee CK, Bustami NA, Tan CK. Acne vulgaris and its association with dietary intake: a Malaysian perspective. Asia Pac J Clin Nutr. 2018;27(5):1141-1145. doi: 10.6133/apjcn.072018.01. PMID 30272862
- [Background] Hanisah A, Omar K, Shah SA. Prevalence of acne and its impact on the quality of life in school-aged adolescents in Malaysia. J Prim Health Care. 2009 Mar;1(1):20-5. PMID 20690482
- [Background] F.B.-B. Yap, The impact of acne vulgaris on the quality of life in Sarawak, Malaysia, Journal of the Saudi Society of Dermatology & Dermatologic Surgery, 16 (2012) 57-60.
- [Background] Lim TH, Badaruddin NSF, Foo SY, Bujang MA, Muniandy P. Prevalence and psychosocial impact of acne vulgaris among high school and university students in Sarawak, Malaysia. Med J Malaysia. 2022 Jul;77(4):446-453. PMID 35902934
- [Background] Loh KC, Chan LC, Phang LF. Perceptions and psychosocial judgement of patients with acne vulgaris. Med J Malaysia. 2020 Jan;75(1):18-23. PMID 32008014
- [Background] J.H. Draize, G. Woodard, H.O. Calvery, Methods for the study of irritation and toxicity of substances applied topically to the skin and mucous membranes, Journal of Pharmacology and Experimental Therapeutics, 82 (1944) 377-390.
- [Background] A.F.M. Hani, A.S. Malik, F.B. Yap, R. Ramli, Segmentation of Acne Vulgaris Lesions, in: Digital Image Computing: Techniques and Applications, Noosa, Queensland Australia, 2008, pp. 335-339.